CLINICAL TRIAL: NCT02754232
Title: Telemedical Training in a Daily Perspective for Chronically Ill COPD Patients: a Cross Sectoral Study
Brief Title: Telemedical Training for Chronically Ill COPD Patients: a Cross Sectoral Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to resource problems in the clinic at University Hospital Odense
Sponsor: Odense University Hospital (Other)
Collaborators: TREFOR (Unknown); CoLab Denmark (Unknown); Region of Southern Denmark (Other); University of Southern Denmark (Other); Danish Lung Association (Other)
Responsible Party: Principal Investigator, Kathrine Rayce, Ph.d. student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT2016
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Physical training; Telemedicine; Daily activities; Cross sectoral
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedical training (Active Comparator): Patients in the intervention group will receive telemedical training 21 times, three times weekly for seven weeks. During the first three weeks the regional physiotherapists will be responsible for the training. Municipal occupational -and physiotherapists will manage the last four weeks' training.
  Interventions: Other: Telemedical training
- The usual training or no training (No Intervention): Patients in the control-group will receive no telemedical training. They will be discharged to the municipal sphere with a rehabilitation plan, where they have the possibility to receive training.

INTERVENTIONS:
Other: Telemedical training — Intervention will involve resistance training and anaerobic training
  Arms: Telemedical training

SUMMARY:
Problem:

Training is an important part of the treatment and rehabilitation of patients with chronic obstructive pulmonary disease (COPD) because training can increase the patient's muscle mass, lead to higher physical performance, reduce difficulties in breathing and hereby increase the patients' capacity to make use of the medical treatment.

Rehabilitation is provided by hospitals training centres/outpatient clinics. However, the transport is too tiring for the patients, which is why they decline taking part in it. This can mean a worsening of their condition and an increase in readmissions.

Solution:

* To develop a better treatment for patients with severe COPD: Telemedical training of patients with COPD in teams.
* To develop a cross-sectoral practice for the telemedical training patients will use, thus decreasing the readmissions of OUH's patients with severe COPD
* To optimize the patient's journey in and across sector borders by using Lean methods.

Perspective:

The study is expected to contribute to improving treatment of severely ill patients with COPD cross-sectorally. The results are expected to contribute to reducing readmissions and raising the level of evidence in telemedical research on training patients with severe COPD. The study's findings may be of use in relation to other patient groups who have difficulties coming to training.

Background:

This research project has its starting point in a pilot project. Its goal was to determine whether severely ill COPD patients could train at home and earlier than normal. Evaluation showed patients found it reassuring to train with the help of the COPD briefcase. They found it increased their physical and mental well-being.

Method:

To gain knowledge of the effect of telemedical training. The patient's strength, daily activity level and quality of life will be measured by conducting a randomized controlled trial including 125 patients - 62 in the intervention group and 62 in the control group.

Qualitative research methods will be used to explore the user perspective concerning patients, family and health professionals. The method is critical psychological practice research.

A Lean method consultant from University Hospital Odense (OUH) will be involved in developing the best clinical pathway for the patients and the professionals.

DETAILED DESCRIPTION:
Project Description:

Problem:

Training is an important part of the treatment and rehabilitation of patients with Chronic Obstructive Pulmonary Disease (COPD) because training can increase the patients' muscle mass, lead to higher physical performance, reduce difficulties in breathing and hereby improve the patient's ability to make use of the medical treatment.

Rehabilitation is provided by hospitals training centres/outpatient clinics. However, the transport is too tiring for the patients, which is why they decline taking part in it. This can mean a worsening of their condition and an increase in readmissions.

Solution:

* To develop a better treatment for patients with severe COPD: Telemedical training of patients with COPD in teams.
* To develop a cross-sectoral practice for the telemedical training patients will use, thus decreasing the readmissions of OUH's patients with severe COPD
* To optimize the patients' journey in and across sector borders by using Lean methods.

The projects relevance for the clinic and target group:

The study is expected to contribute to improving the treatment of severely ill patients with COPD cross-sectorally by generating knowledge for the physical and occupational therapists' practice. The results are expected to contribute to reducing readmissions and raising the level of evidence in telemedical research on training patients with severe COPD.

The study includes patients with severe COPD in Odense and Svendborg. It is anticipated that similar patient groups with similar difficulties, nationally as well as internationally, will benefit from the findings.

Background:

More than 430.000 people in Denmark have Chronic Obstructive Pulmonary Disease (COPD) (Hansen et al., 2008). Characteristic for COPD is respiratory tract obstruction, which is not completely reversible and worsens as time passes. Complications of COPD are: loss of muscle mass, weight loss and an increasing social isolation (The National Board of Health, 2007).

It is well documented that a systematic individually composed rehabilitation program, including training, has an effect on patients' functional level and quality of life (National board of Health, 2007). Early rehabilitation after hospitalization may break the vicious circle, which can arise for patients with COPD. In this cycle, hospitalization can entail inactivity and loss of muscular strength, thus increasing the risk of new aggravations with re-admittance to hospital as a result (National board of Health, 2014). In addition, at this time no studies examine the effect of training on daily activities (ibid).

To offer these severely ill patients rehabilitation is a regional task. However, the patients with severe COPD often decline training, as the transport to and from hospital is too exhausting for them. The result is no training for this group. The same dilemma exists in other countries (Burkow et al., 2013). Inactivity can mean stagnation in daily life, which affects functioning (Williams et al., 2011) for both patients and their families (Wong et al., 2005) Patients with COPD, who cannot take part in the usual rehabilitation program due to the degree of their illness, are now recommended to take part in strength training as a replacement. The recommendation is based solely on consensus of good clinical practice. Research is lacking (National Board of Health, 2014).

Few studies examine telemedicine, COPD and supervised training. Two studies with supervised team training for, among others, patients with COPD showed great patient satisfaction and an increased experience of social support (Nield and Hoo, 2012, Burkow et al., 2013). One of the studies showed a significantly decreased occurrence of dyspnoea in the intervention group (Nield and Hoo, 2012).

In 2010-2012 OUH did a feasibility study in an attempt to develop a training program for patients with severe or very severe COPD who reject the established rehabilitation program at the hospital. The study, which encompassed 50 patients in a year, tested and developed an early effort using an individually tailored home-training program based on telemedical training.

The results showed potential in relation to previous telemedical training of patients with COPD. Considering the scanty knowledge in the field, a contribution to produce knowledge of greater variation is relevant.

Project type:

An randomised controlled Study (RCT) is needed to reveal the effect of telemedical training and muscle strength related to doing every day chores and to see how this affects their daily activities and quality of life.

The RCT study:

Aim:

The aim is to study the effect of telemedical training on activities of daily living, quality of life and physical performance in patients with severe or very severe COPD.

Hypotheses:

This study is designed to assess the hypothesis that patients with severe or very severe COPD, who have thanked no to training at the hospital, receiving telemedical training will experience greater satisfaction doing daily activities, increase their quality of life and increase their physical performance than patients who do not receive telemedical training.

Place and project participants:

Patients who take part in the study have been admitted to OUH because of a worsening of their COPD. The criteria for inclusion and exclusion criteria will be submitted elsewhere.

Design and method:

The project participants are included consecutively in the intervention group or the control group for two years. A power calculation shows the study can, with a random sampling size of 100 patients, 50 in each group, show a difference of 2,7 seconds in FTSST(Stand up - sit down five times). The strength is set to 80 %. The calculation is based on a standard deviation of 4,8 for FTSST and a 5 % to-sided significance level. If a dropout rate of 20 % is allowed for, it will mean that 128 persons must be included.

The patients are randomized to the intervention group or the control group by baseline after an informed consent. Measurements are made at baseline, post-intervention and follow-up, which are 3 and 6 months after post-intervention.

Patients in the intervention group will receive telemedical training in teams of up to 4, 21 times, three times weekly for seven weeks. During the first three weeks the regional physiotherapists will be responsible for the training. Municipal occupational -and physiotherapists will manage the last four weeks' training.

Patients in the control-group will receive no training as they have refused the offer. They will be discharged to the municipal sphere with a rehabilitation plan.

Data generation method:

Function tests and questionnaires will be included in the quantitative study of the telemedicial training's importance for physical ability, daily activities and health related quality of life for patients with severe or very severe COPD.

Outcome measures will be submitted elsewhere. The following parameters describe the participating patient group: Sex, age, civil status, socio - economic status, Body Mass Index (BMI), forced expiratory volume in one 1 second (FEV1) of expected value, FEV1 / forced vital capacity (FVC), Medical Research Council Breathlessness Scale (MRC- dyspnea score), oxygen treatment in the home, treatment with atomizer, the usual inhaled COPD treatment (grouped), oral prednisolone treatment, home care, use of tobacco.

Whether telemedical training has an effect on readmissions for patients with COPD will be examined by comparing the number of admissions for the intervention group and the control group. Data will be requisitioned from the Region's IT.

Analysis:

The data will be continuously keyed into an Access database. Calculation of the analysis will be done using the software program STATA (abbreviation of Statistic and Data). The data will be analyzed according to the principle 'intention to treat'. The level of significance α will be placed at 0,05 and power β = 0,8. Descriptive statistics and regression analysis will be used.

Ethical considerations:

The patients will be informed of the project's goal, form and content both orally and in written form and that participation is voluntary. Written consent must be had before inclusion. Participants will be informed that they can leave the study at any time. The project leader will file inclusion numbers and corresponding personal data securely according to the applicable rules. The project is registered and approved of by The Danish Data Protection Agency and the Danish Council of Ethics.

Documentation of results, knowledge sharing and distribution:

Three articles will be published in relevant international peer-reviewed journals. The Danish Lung Association will be continuously informed of the study's status. The results will be distributed to national and international conferences, and studies abroad. These include health professional forums during the Ph.D. study - depending on the results of the study.

Database:

Data from the project will be stored via Odense Patient Explorative Network (OPEN)- more specifically Redcap as the data management system. Redcap is approved of by God Clinical practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* patients with severe and very severe COPD, that is FEV1/FVC under 0,7, FEV1 under 50 % of the expected value and grade three and above on the Medical Research Council Dyspnoea Scale (MRC- Dyspnoea Scale).
* The patients have rejected OUH's offer of training at the hospital.
* The patients must be mobile enough to complete the training.
* The patients are motivated to participate in individual adjusted telemedical training in teams.
* The patients have at the same time been offered Telemedical consultations by a nurse
* The patients biggest problem concerning physical activity has to be their shortness of breath
* The patients live in either Svendborg or Odense

Exclusion Criteria:

* patients with lacking ability to communicate via telephone and/or computer screen, severe kidney insufficiency or cardiac insufficiency, saturation less than 88 % and possibly malignant changes in lung(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The Stand up - sit down five times test (FTSST) | 7 weeks
  The FTSST test (Stand up - sit down five times) is a function test, which measures lower body strength. It gives a picture of the ability to get up from a chair, which is a daily activity. The smallest relevant change is 2,7 seconds (Reuben and Siu, 1990). Whether patients continue rehabilitation training in the municipal sphere, after telemedical training is completed is also noted.

SECONDARY OUTCOMES:
The Clinical COPD Questionnaire (CCQ) | 3 and 7 weeks, 3 and 6 months
  The Clinical COPD Questionnaire (CCQ) is a validated questionnaire, measuring the health status for patients with COPD by using a standardized self-administered questionnaire about COPD. CCQ is useful for comparing measurements of health status at group level. In addition for quantifying changes in health after treatment and correlating with COPD Assesment Test (CAT) and Saint George's Respiratory Questionnaire (SGRQ)
The Activities of Daily Living Questionnaire (ADL - Q) | 7 weeks, 3 and 6 months
  ADL - Q is a questionnaire, completed by the patient that measures the individual's perception of their own abilities to carry out daily activities
Physical Activity Scale | 3 and 7 weeks, 3 and 6 months
  The Physical Activity Scale is a validated questionnaire, completed by the patient that measures the extent of a participant's physical activity on an average 24 hour period
The Stand up - sit down five times test (FTSST) | 3 weeks, 3 and 6 months
  The FTSST test (Stand up - sit down five times) is a function test, which measures lower body strength. It gives a picture of the ability to get up from a chair, which is a daily activity. The smallest relevant change is 2,7 seconds (Reuben and Siu, 1990). Whether patients continue rehabilitation training in the municipal sphere, after telemedical training is completed is also noted.
Readmissions | 3 and 6 months
  Whether telemedical training has an effect on readmissions for patients with COPD will be examined by comparing the number of admissions for the intervention group and the control group. Data will be requisitioned from the Region's IT.
Walking distance | 3 and 7 weeks, 3 and 6 months
  The participants will be asked if they can walk 300 meters. This has shown to be a good clinical determinants of a poor 6-min walking distance (<350 m) in patients with COPD (Spruit M. et al 2009)
European Quality of Life-5 Dimensions (EQ5D) | 3 and 7 weeks, 3 and 6 months
  EQ5D is a validated questionaire, developed to estimate health status (Brooks, 1996)

OTHER OUTCOMES:
Participation in municipial or private training | 3 and 7 weeks, 3 and 6 months
  We are interested in knowing whether the patients in the intervention or control group participate in (other) training. there are no questionaire connected to this question, we simply ask the patients.
The total cost of treatment compared with effectiveness | 7 weeks,3 and 6 months
  The cost-effective analysis estimates the total cost of the intervention (equipment and use of staff per patient) and the economic advantages such as a decline in readmissions. The total net costs are compared to the clinical changes.
System Usability Scale (SUS) | 7 weeks
  A questionaire used in economic evaluation for estimating the satisfaction and safety of the users of the technology

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Kidholm, Ass professor, Study Director — University Hospital Odense